CLINICAL TRIAL: NCT01313052
Title: Forensic Assertive Community Treatment: An Emerging Model of Service Delivery
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven Lamberti, Professor, Department of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R34MH078003-03 (NIH); 5R34MH078003-03 (NIH)
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Psychotic Disorders
Keywords: Psychotic; Criminal
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forensic Assertive Community Treatment (FACT) (Experimental): Individuals in this arm will receive the services of an Assertive Community Treatment team and close supervision of a judge trained in the FACT model.
  Interventions: Behavioral: Forensic Assertive Community Treatment (FACT)
- Enhanced Treatment as Usual (Active Comparator): Individuals in this arm of the study will receive an expedited appointment at a clinic specializing in the treatment of psychotic disorders. These individuals will receive the services of a therapist, psychiatrist, and case manager.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Forensic Assertive Community Treatment (FACT) — Individuals in this arm will receive the services of an Assertive Community Treatment team and close supervision of a judge trained in the FACT model.
  Arms: Forensic Assertive Community Treatment (FACT)
Behavioral: Enhanced Treatment as Usual — Individuals in this arm of the study will receive an expedited appointment at a clinic specializing in the treatment of psychotic disorders. These individuals will receive the services of a therapist, psychiatrist, and case manager.
  Arms: Enhanced Treatment as Usual

SUMMARY:
The FACT model (ACT + legal leverage in the form of judicial monitoring) will be compared to enhanced outpatient treatment (close outpatient follow-up without judicial monitoring). Seventy adults with psychotic disorders in Monroe County who are convicted of a misdemeanor will be randomly assigned to each treatment group and followed for 12 months. Primary outcomes will include criminal justice and mental health service utilization rates, treatment adherence, psychiatric symptoms, substance abuse, homelessness, perceived coercion, and consumer satisfaction. Service utilization outcomes will be tracked using established mental health and criminal justice databases.

Hypotheses are:

1. FACT (ACT plus judicial monitoring) will have a greater effect than enhanced TAU in promoting treatment adherence among high-risk adults with psychotic disorders.
2. FACT (ACT plus judicial monitoring) will have a greater effect than enhanced TAU in preventing arrest, incarceration, emergency department and inpatient hospital use among high-risk adults with psychotic disorders.

DETAILED DESCRIPTION:
FACT (Forensic Assertive Community Treatment) is an adaptation of the Assertive Community Treatment (ACT) model that addresses a significant gap in our service delivery systems by targeting the interface between mental health and criminal justice services. ACT was originally developed to engage severely mentally ill adults in outpatient psychiatric treatment through the use of assertive outreach and comprehensive services. FACT adds legal leverage in the form of judicial monitoring to ACT, which is comprehensive, high intensity, mobile, psychiatric treatment.

The FACT model (ACT + legal leverage in the form of judicial monitoring) will be compared to enhanced outpatient treatment (close outpatient follow-up without judicial monitoring). Seventy adults with psychotic disorders in Monroe County who are convicted of a misdemeanor will be randomly assigned to each treatment group and followed for 12 months. Primary outcomes will include criminal justice and mental health service utilization rates, treatment adherence, psychiatric symptoms, substance abuse, and homelessness. Service utilization outcomes will be tracked using established mental health and criminal justice databases.

Hypotheses are:

1. FACT (ACT plus judicial monitoring) will have a greater effect than enhanced TAU in promoting treatment adherence among high-risk adults with psychotic disorders.
2. FACT (ACT plus judicial monitoring) will have a greater effect than enhanced TAU in preventing arrest, incarceration, emergency department and inpatient hospital use among high-risk adults with psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with any psychotic disorder such as Schizophrenia, Schizoaffective Disorder, Bipolar Disorder with Psychotic Features, Depressive Disorder with Psychotic Features, and Psychotic Disorder, Not Otherwise Specified.
* Individuals currently facing misdemeanor or violation charges who have not yet been sentenced.

Exclusion Criteria:

* Individuals do not have or cannot be diagnosed with a psychotic disorder.
* Individuals currently facing felony charges
* Individuals currently involved in any type of legal leverage including probation, parole, drug or mental health court supervision, Assisted Outpatient Treatment, or Criminal Procedure Law status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Jail Recidivism | For the one year subjects are in the study.
  The study will measure number of arrests, number of incarcerations, and total number of jail and/or prison days in the time frame described above.
Mental Health Service Utilization | For the one year subjects are in the study.
  The study will measure number of hospitalizations, number of hospital days, number of emergency room visits, number of outpatient mental health visits as primary outcome measures, and treatment appointment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: J Steven Lamberti, MD, Principal Investigator — University of Rochester
Locations (1):
- Monroe County Jail, Rochester, New York, United States

REFERENCES:
- [Background] Lamberti JS, Deem A, Weisman RL, LaDuke C. The role of probation in forensic assertive community treatment. Psychiatr Serv. 2011 Apr;62(4):418-21. doi: 10.1176/ps.62.4.pss6204_0418. PMID 21459994
- [Background] Lamberti, J., & Weisman, R. (2010). Forensic assertive community treatment: Origins, current practice, and future directions. In H. Dlugacz (Ed.), Reentry Planning for Offenders With Mental Disorders (1 ed., Vol. 1, pp. 145-169). Kingston, NJ: Civic Research Institute.
- [Result] Lamberti, JS. (2011). Legal Leverage in the Treatment of Adults With Severe Mental Illness, in Workplace Violence in Mental Health and General Health Care Settings. Pages 225 - 236. M. Privitera, editor. Jones and Bartlett, Pages 225-236.